CLINICAL TRIAL: NCT06250465
Title: AGMT Austrian CLL (Chronic Lymphocytic Leukemia) Registry
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_CLL-Reg
Record Dates: First submitted 2022-08-25; First posted 2024-02-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — The CLL registry will be accompanied by an optional biobanking program. Sample collection will be limited to patients that have signed an additional biobanking IC. The samples are taken as part of the clinical routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
For until very recently CLL has been considered an uncurable disease, with the only few exceptions of a part of patients capable of undergoing and successfully standing allogeneic stem cell transplant. However, the introduction of chemoimmunotherapy in particular the FCR (fludarabine, cyclophosphamide, rituximab) regimen has established a relevant population of IgVH mutated patients, who remain relapse-free for up to 10 years with a clear plateau at this level. However, for the largest proportion of all CLL patients the disease is still associated with a reduction in life expectancy as compared to a matched population.

The field has made further substantial progress by the introduction of BTK inhibitors and Bcl2 inhibitors, novel antibodies as well as by the understanding of the role of minimal residual disease (MRD), mutations and their clonal evolution over time as risk factors and factors governing the kind and duration of therapy.

Due to the limited follow up of frontline therapy trials using novel drugs, it is not yet clear, what the long-term results with many of the new drugs will be. Particularly, long-term PFS, the potential for cure and the long-term safety issues remain relevant parameters requiring examination, as are infections, interactions with other drugs or quality of life issues.

CLL has not been systematically assessed in Austria to date. This medical registry of the AGMT is thus the first Austrian-wide standardized documentation of this disease.

DETAILED DESCRIPTION:
This registry is designed as multicenter observational cohort of patients with CLL. Patient medical, testing and treatment information will be obtained through extraction of data from existing patient medical charts. Longitudinal follow-up data, including survival and tumor progression, will also be extracted from patient medical charts. This patient follow-up data will be obtained until patient death or loss to follow-up.

For documentation in the registry, no further diagnostic or therapeutic measures are required than those already necessary in general. Participation in the registry must not interfere with treatment routines. Only routine data, which has already been recorded in the patient's medical chart, is transferred to the electronic Case Report Forms. To maintain patient confidentiality, each patient will be assigned a unique patient identifying number upon enrollment; this number will accompany the patient's medical and other registry information throughout the lifetime of the registry.

A written consent must be obtained prior to the input of data. No informed consent is required from deceased patients.

ELIGIBILITY:
Inclusion Criteria:

* The registry will include patients ≥ 18 years with CLL.

Exclusion Criteria:

* There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Austrian sites that treat patients in this indication will be invited to participate in this registry.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
General Characteristics | 7 years
  To describe general characteristics of CLL patients
Genetic Profiling | 7 years
  To describe genetic risk profiles
Proportion of CLL patients in Austria that require treatment | 7 years
  To describe the proportion of CLL patients in Austria that require treatment
Number of patients with concomitant diseases | 7 years
  To describe concomitant diseases at diagnosis of CLL
Number and type of treatment | 7 years
  To describe type and duration of treatment of CLL. Number of patients per treatment, number of treatments per patient.
Patient Outcome | 7 years
  To describe patient outcome (complete response, partial response...) in relation to the type of treatment administered.
Toxicities | 7 years
  To describe toxicity with a focus on infections, cardiotoxicity, nephrotoxicity, bleeding, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — Department of internal Medicine III, Paracelsus Medical University Salzburg, Austria
Locations (9):
- Austria (9):
  - Landeskrankenhaus Feldkirch, Innere Med. II, Interne E, Feldkirch
  - Univ.-Klinik für Innere Medizin V, Hämatologie/Onkologie LKH-Innsbruck / Universitätskliniken, Innsbruck
  - A.ö. Bezirkskrankenhaus Kufstein, Innere Medizin / Hämatologie / Onkologie, Kufstein
  - KUK Linz: Klinik für Interne 3 - Schwerpunkt Hämatologie und Onkologie, Linz
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern; Interne I: Medizinische Onkologie und Hämatologie, Linz
  - Ordensklinikum Linz GmbH, Elisabethinen, I. Interne Abteilung Hämato-Onkologie, Linz
  - UK Salzburg, LKH: Universitätsklinik für Innere Medizin III, Salzburg
  - Univ.-Klinikum St. Pölten, Innere Medizin 1, Sankt Pölten
  - Klinikum Wels-Grieskirchen, Abteilung für Innere Medizin IV, Wels

IPD SHARING:
Plan to Share IPD: No